CLINICAL TRIAL: NCT05793359
Title: Comparison of the Efficacy of Two Different Glucocorticoid Regimens for Treatment of Active Moderate-to-severe Graves' Orbitopathy
Brief Title: Comparison of the Effectiveness of Two Glucocorticoid Regimens for Treatment of Graves' Orbitopathy
Status: Completed | Type: Observational
Sponsor: Medical University of Sofia (Other)
Responsible Party: Principal Investigator, Mariya Stoynova, Principal investigator, Medical University of Sofia
Other Study IDs: 21A /25.07.2017
Record Dates: First submitted 2023-03-07; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Graves Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Methylprednisolone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Modified monthly regimen: Treatment with 3 pulses of 3 infusions of 500 mg methylprednisolone on 3 consecutive months with intramuscular administration of 125 mg methylprednisolone per week between the pulses. Additional low dose peroral treatment after completion of the pulses.
  Interventions: Drug: Methylprednisolone
- Weekly regimen: Treatment with 6 infusions of 500 mg methylprednisolone during the first 6 weeks, followed by 6 infusions of 250 mg methylprednisolone during the next 6 weeks.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — methylprednisolone applied as intravenous infusions or intramuscularly
  Other Names: Urbason

SUMMARY:
The goal of this interventional study is to compare the effectiveness of two different glucocorticoid regimens for treatment of active moderate-to-severe Graves' orbitopathy. The main questions it aims to answer are:

1. Are the two glucocorticoid regimens similarly effective?
2. Do the two glucocorticoid regimens have similar safety profile? The patients involved are treated with one of the two glucocorticoid regimens. Their ocular status, therapeutic response and quality of life reassessed during the treatment, at its end, and 3 month later.

DETAILED DESCRIPTION:
Systemic glucocorticoids are the mainstay of treatment for active moderate-to-severe Graves' orbitopathy. However, there are a number of different glucocorticoid regimens with different total dosage, schemes of administration and duration. The goal of this interventional study is to compare the effectiveness of two different glucocorticoid regimens for treatment of active moderate-to-severe Graves' orbitopathy. The main questions it aims to answer are:

1. Are the two glucocorticoid regimens similarly effective?
2. Do the two glucocorticoid regimens have similar safety profile? The patients involved are treated with one of the two glucocorticoid regimens. The first group is treated with modified monthly regimen, including 3 pulses of 3 infusions of 500 mg methylprednisolone administered in three consecutive months, with application of 125 mg methylprednisolone intramuscularly once per week between the pulses. Total cumulative dose - 5.5. g., duration - 3 months. After completion of the venous infusions, a low dose peroral glucocorticoid therapy is prescribed for the next 3 months. The second group is treated with weekly glucocorticoid regimen: 6 infusions of 500 mg methylprednisolone during the first 6 weeks followed by 6 infusions of 250 mg methylprednisolone during the next 6 weeks. Total cumulative dose - 4.5 g., duration - 3 months. Patients' ocular status and therapeutic response are assessed at 1st, 3rd and 6th months; quality of life - at 3rd and 6th month.

ELIGIBILITY:
Inclusion Criteria:

* Active moderate-to-severe Graves' orbitopathy
* Without previous treatment with glucocorticoids or orbital radiotherapy
* Euthyroid state

Exclusion Criteria:

* Uncontrolled hyper- or hypothyroidism
* Previously treated Graves' orbitopathy
* Mild or sight-threatening form of Graves' orbitopathy
* Inactive moderate-to-severe Graves' orbitopathy
* Contraindications for glucocorticoid treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixty-two patients with untreated active moderate-to-severe Graves' orbitopathy in euthyroid state under treatment.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Comparison of the changes in the overall therapeutic response assessed using Bartalena's criteria during the treatment with the two glucocorticoid regimens | 6 months
  Comparison of the changes in the overall therapeutic response assessed using Bartalena's criteria and classified as full, partial and no response during the treatment with the two glucocorticoid regimens
Comparison of the changes in clinical activity score, assessed using a 7- or 10-point scale and expressed in points during the treatment with the two glucocorticoid regimens | 6 months
  Comparison of the changes in clinical activity score, assessed using a 7-point scale at baseline or 10-point scale during the follow-up and expressed in points as recommended by European Thyroid Association and European Group on Graves' orbitopathy during the treatment with the two glucocorticoid regimens
Comparison of the changes in lid aperture expressed in mm during the treatment with the two glucocorticoid regimens | 6 months
  Comparison of the changes in lid aperture measured by ruler and expressed in mm during the treatment with the two glucocorticoid regimens
Comparison of the changes in proptosis expressed in mm during the treatment with the two glucocorticoid regimens | 6 months
  Comparison of the changes in proptosis measured by Hertel's exophthalmometer and expressed in mm during the treatment with the two glucocorticoid regimens
Comparison of the changes in visual acuity expressed in decimals during the treatment with the two glucocorticoid regimens | 6 months
  Comparison of the changes in visual acuity measured by Snellen chart and expressed in decimals during the treatment with the two glucocorticoid regimens
Comparison of the changes in diplopia assessed using Gorman's classification system during the treatment with the two glucocorticoid regimens | 6 months
  Comparison of the changes in diplopia assessed using Gorman's classification system and classified as gr. 0 absent, gr. I intermittent, gr. II inconstant, gr. III constant during the treatment with the two glucocorticoid regimens
Comparison of the changes in soft tissue involvement evaluated using the colour atlas proposed by European Group on Graves' orbitopathy during the treatment with the two glucocorticoid regimens | 6 months
  Comparison of the changes in soft tissue involvement evaluated using the colour atlas proposed by European Group on Graves' orbitopathy and categorized as gr. 0-I absent or mild, gr. II-III moderate or severe during the treatment with the two glucocorticoid regimens
Comparison of the changes in subjective symptoms whose severity was reported by patients themselves using subjective scale during the treatment with the two glucocorticoid regimens | 6 months
  Comparison of the changes in subjective symptoms whose severity was reported by patients themselves and were graded as 0-I absent or mild, gr. II-III moderate or severe during the treatment with the two glucocorticoid regimens
Comparison of the changes in quality of life assessed by disease-specific questionnaire recommended by European Group on Graves' orbitopathy (GO-QoL) аnd expressed as percentages during the treatment with the two glucocorticoid regimens | 6 months
  Comparison of the changes in quality of life during the treatment with the two glucocorticoid regimens assessed by disease-specific questionnaire recommended by European Group on Graves' orbitopathy (GO-QoL) аnd expressed as percentages, which includes two subscales - one evaluating the impact of Graves' orbitopathy on patients' visual functioning (QoL-VF) and the other related to the changes of physical appearance as a result of the disease (QoL-AP)
Incidence of treatment-emerged adverse events in the two glucocorticoid regimens groups | 6 months
  Number and type of adverse reactions in the study groups reported by patients themselves or found by the laboratory tests or during clinical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Mariya D Stoynova, PhD, Principal Investigator — Medical University of Sofia: Medicinski universitet-Sofia
Locations (1):
- University Hospital of Endocrinology, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stoynova MA, Shinkov AD, Dimitrova ID, Yankova IA, Kovatcheva RD. Comparison of the efficacy of two different glucocorticoid regimens for treatment of active moderate-to-severe Graves' orbitopathy. Int Ophthalmol. 2023 Dec;43(12):4747-4757. doi: 10.1007/s10792-023-02875-z. Epub 2023 Sep 12. PMID 37698660